CLINICAL TRIAL: NCT02548793
Title: CPR Education for Families of Cardiac Patients Before Hospital Discharge
Brief Title: CPR Education Via a Mobile Application Compared to VSI Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 822593
Record Dates: First submitted 2015-08-31; First posted 2015-09-14 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Risk Factors; Coronary Disease; Cardiac Arrest
Keywords: Cardiac Arrest; CPR; Family-centered Care; Health Literacy; Health Education; Education Dissemination
MeSH Terms: conditions — Coronary Disease; Heart Arrest; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSI Kit (Active Comparator): Education: CPR Training using the CPR Anytime VSI Kit Individuals will learn chest-compression only CPR (no rescue breaths) using the American Heart Association's Family and Friends CPR Anytime Kit. Subjects will undergo training in-hospital and will be encouraged to take the kit home to share with their family members and friends.
  Interventions: Other: Education: CPR Training using the CPR Anytime VSI Kit
- Mobile Application (Experimental): Education: CPR Training via Mobile App Individuals will learn chest-compression only CPR (no rescue breaths) using a newly developed mobile training application.
  Interventions: Other: Education: CPR Training via Mobile App

INTERVENTIONS:
Other: Education: CPR Training via Mobile App — Using a mobile app to train users on chest-compression only CPR. Subjects will be encouraged to share the app with family and friends.
  Other Names: CPR Training Cellphone App
  Arms: Mobile Application
Other: Education: CPR Training using the CPR Anytime VSI Kit — Subjects will be trained using the American Heart Association's Family and Friends CPR Anytime Kit. Subjects will undergo training in-hospital and will be encouraged to take the kit home to share with their family members and friends.
  Other Names: Family and Friends CPR Anytime; American Heart Association Family and Friends CPR Anytime; CPR Anytime Video Self Instruction (VSI)
  Arms: VSI Kit

SUMMARY:
Prompt delivery of cardiopulmonary resuscitation (CPR) is a crucial determinant of survival for many victims of sudden cardiac arrest (SCA), yet bystander CPR is provided in less than one third of witnessed SCA events. A number of barriers to bystander CPR training have been identified including time and cost of the training course. Since the large majority of arrest events occur in the home environment, studies have suggested that providing CPR training to family members of hospitalized cardiac patients may serve as a useful approach to address an environment in which bystander CPR is frequently not provided. Utilizing an existing in-hospital program to train adult family members, the investigators will assess the skills of those who learn CPR through two different educational methods: a mobile app and video self-instruction (VSI).

DETAILED DESCRIPTION:
The long term goal of the investigators work is to implement real world CPR training strategies that match training locales with at-risk populations, maximize resuscitation skill retention, and promote willingness to act. To accomplish this, the investigators will empower stakeholders at the University of Pennsylvania Health System (UPHS) and local area hospitals to develop local implementation approaches, using either volunteer hospital personnel or paid research assistants as training proctors. These stakeholders will be studied as a research subset. The training proctors will educate family members or friends of patients at risk for cardiac arrest using a mobile application "app" or VSI kit (RCT), and empower them with the lifesaving skill of CPR. The investigators will follow up with the study subjects and conduct CPR skills tests 6 to 12 months from the time of training to assess whether the subjects retained their skills or if they had an opportunity to use the skills that they learned. The investigators will also gather information on how the subjects would like to be encouraged to practice their skills. The investigators will send a reminder notification every two months following training, to encourage subjects to refresh their training skills. At the follow-up skills test at 6 to 12 months, the investigators will administer a survey to assess whether the prompting encouraged the subjects to practice their skills. Additionally the investigators will encourage the individuals trained in-hospital to share the kit or mobile app with others. The investigators will follow-up with those who are identified as secondary trainees to assess the environment in which secondary training took place.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be present with their family member at the hospital
* The family member must be at high risk for cardiac arrest (CA), including:
* previous myocardial infarction (MI)
* previous CA
* history of diabetes
* history of high cholesterol
* history of high blood pressure
* This includes subjects with family members being discharged from the Cardiac Intermediate Care Unit (CICU), Telemetry units, ICU, Cardiac Care Unit (CCU), cardiology clinics, or physicians office within the participating hospitals/health systems

Exclusion Criteria:

* Volunteers and subjects must be 18 years of age or older
* Individual must be fit and able to perform moderate physical activity
* Volunteers must be English speaking and/or Spanish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1679 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Chest compression depth | 6 months
  Depth of chest compression performed by the subject, recorded using the Laerdal SimPad®. This metric will be measured in millimeters (mm). This outcome measure will be collected by research coordinators during 6-month in-home follow-up visits.
Chest compression rate | 6 months
  Rate of chest compressions performed by the subject, recorded using the Laerdal SimPad®. This metric will be measured as the number of compressions performed in a 2 minute window. This outcome measure will be collected by research coordinators during 6-month in-home follow-up visits.

SECONDARY OUTCOMES:
Secondary CPR training rates | 6 months
  Calculate the number of secondary trainees based on study participant self-reporting (via survey) collected during the 6-month follow-up.
Incidence of bystander CPR provided by subjects | 6-12 months
  Using 6 month and 12 month follow-up surveys, subjects will be asked if they had an opportunity to use their CPR skills in a real-life situation and whether or not they performed CPR in the aforementioned situation.

OTHER OUTCOMES:
Qualitative analysis of patient's perspective of the family member's receiving hands-only CPR training using semi-structured | 6-12 months
  Using semi-structured interviews, we will evaluate the impact that CPR training of the patient's family may have on the patient's sense of independence and self-care post-discharge. Analysis will be based on the grounded theory. A working set of thematic codes will be identified and applied to all interview transcriptions using NVivo10. Thematic domains from this descriptive aim will help inform future understanding of the cardiac patient's psychological well-being and preparedness around cardiac disease as well as thoughts towards CPR training.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Abella, MD, MPhil, Principal Investigator — University of Pennsylvania
Locations (7):
- United States (7):
  - Cooper University Hospital, Camden, New Jersey
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Crozer-Keystone Health System, Upland, Pennsylvania
  - The Chester County Hospital and Health System, West Chester, Pennsylvania

REFERENCES:
- [Background] Blewer AL, Leary M, Decker CS, Andersen JC, Fredericks AC, Bobrow BJ, Abella BS. Cardiopulmonary resuscitation training of family members before hospital discharge using video self-instruction: a feasibility trial. J Hosp Med. 2011 Sep;6(7):428-32. doi: 10.1002/jhm.847. Epub 2010 Nov 8. PMID 21916007
- [Background] Blewer AL, Leary M, Esposito EC, Gonzalez M, Riegel B, Bobrow BJ, Abella BS. Continuous chest compression cardiopulmonary resuscitation training promotes rescuer self-confidence and increased secondary training: a hospital-based randomized controlled trial*. Crit Care Med. 2012 Mar;40(3):787-92. doi: 10.1097/CCM.0b013e318236f2ca. PMID 22080629
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Background] Rea TD, Helbock M, Perry S, Garcia M, Cloyd D, Becker L, Eisenberg M. Increasing use of cardiopulmonary resuscitation during out-of-hospital ventricular fibrillation arrest: survival implications of guideline changes. Circulation. 2006 Dec 19;114(25):2760-5. doi: 10.1161/CIRCULATIONAHA.106.654715. Epub 2006 Dec 11. PMID 17159062
- [Background] Stiell IG, Wells GA, Field B, Spaite DW, Nesbitt LP, De Maio VJ, Nichol G, Cousineau D, Blackburn J, Munkley D, Luinstra-Toohey L, Campeau T, Dagnone E, Lyver M; Ontario Prehospital Advanced Life Support Study Group. Advanced cardiac life support in out-of-hospital cardiac arrest. N Engl J Med. 2004 Aug 12;351(7):647-56. doi: 10.1056/NEJMoa040325. PMID 15306666
- [Background] Bagai A, McNally BF, Al-Khatib SM, Myers JB, Kim S, Karlsson L, Torp-Pedersen C, Wissenberg M, van Diepen S, Fosbol EL, Monk L, Abella BS, Granger CB, Jollis JG. Temporal differences in out-of-hospital cardiac arrest incidence and survival. Circulation. 2013 Dec 17;128(24):2595-602. doi: 10.1161/CIRCULATIONAHA.113.004164. Epub 2013 Sep 17. PMID 24045044
- [Background] Cobb LA, Fahrenbruch CE, Walsh TR, Copass MK, Olsufka M, Breskin M, Hallstrom AP. Influence of cardiopulmonary resuscitation prior to defibrillation in patients with out-of-hospital ventricular fibrillation. JAMA. 1999 Apr 7;281(13):1182-8. doi: 10.1001/jama.281.13.1182. PMID 10199427
- [Background] Holmberg M, Holmberg S, Herlitz J; Swedish Cardiac Arrest Registry. Factors modifying the effect of bystander cardiopulmonary resuscitation on survival in out-of-hospital cardiac arrest patients in Sweden. Eur Heart J. 2001 Mar;22(6):511-9. doi: 10.1053/euhj.2000.2421. PMID 11320981
- [Background] Iwami T, Kawamura T, Hiraide A, Berg RA, Hayashi Y, Nishiuchi T, Kajino K, Yonemoto N, Yukioka H, Sugimoto H, Kakuchi H, Sase K, Yokoyama H, Nonogi H. Effectiveness of bystander-initiated cardiac-only resuscitation for patients with out-of-hospital cardiac arrest. Circulation. 2007 Dec 18;116(25):2900-7. doi: 10.1161/CIRCULATIONAHA.107.723411. Epub 2007 Dec 10. PMID 18071072
- [Background] Anderson ML, Cox M, Al-Khatib SM, Nichol G, Thomas KL, Chan PS, Saha-Chaudhuri P, Fosbol EL, Eigel B, Clendenen B, Peterson ED. Rates of cardiopulmonary resuscitation training in the United States. JAMA Intern Med. 2014 Feb 1;174(2):194-201. doi: 10.1001/jamainternmed.2013.11320. PMID 24247329
- [Background] Nichol G, Thomas E, Callaway CW, Hedges J, Powell JL, Aufderheide TP, Rea T, Lowe R, Brown T, Dreyer J, Davis D, Idris A, Stiell I; Resuscitation Outcomes Consortium Investigators. Regional variation in out-of-hospital cardiac arrest incidence and outcome. JAMA. 2008 Sep 24;300(12):1423-31. doi: 10.1001/jama.300.12.1423. PMID 18812533
- [Background] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Background] Abella BS, Aufderheide TP, Eigel B, Hickey RW, Longstreth WT Jr, Nadkarni V, Nichol G, Sayre MR, Sommargren CE, Hazinski MF; American Heart Association. Reducing barriers for implementation of bystander-initiated cardiopulmonary resuscitation: a scientific statement from the American Heart Association for healthcare providers, policymakers, and community leaders regarding the effectiveness of cardiopulmonary resuscitation. Circulation. 2008 Feb 5;117(5):704-9. doi: 10.1161/CIRCULATIONAHA.107.188486. Epub 2008 Jan 14. No abstract available. PMID 18195177
- [Background] Cho GC, Sohn YD, Kang KH, Lee WW, Lim KS, Kim W, Oh BJ, Choi DH, Yeom SR, Lim H. The effect of basic life support education on laypersons' willingness in performing bystander hands only cardiopulmonary resuscitation. Resuscitation. 2010 Jun;81(6):691-4. doi: 10.1016/j.resuscitation.2010.02.021. Epub 2010 Mar 26. PMID 20347208
- [Background] Swor R, Compton S. Estimating cost-effectiveness of mass cardiopulmonary resuscitation training strategies to improve survival from cardiac arrest in private locations. Prehosp Emerg Care. 2004 Oct-Dec;8(4):420-3. doi: 10.1016/j.prehos.2004.06.012. PMID 15626005
- [Background] Brennan RT, Braslow A. Are we training the right people yet? A survey of participants in public cardiopulmonary resuscitation classes. Resuscitation. 1998 Apr;37(1):21-5. doi: 10.1016/s0300-9572(98)00026-4. PMID 9667334
- [Background] Free C, Phillips G, Watson L, Galli L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technologies to improve health care service delivery processes: a systematic review and meta-analysis. PLoS Med. 2013;10(1):e1001363. doi: 10.1371/journal.pmed.1001363. Epub 2013 Jan 15. PMID 23458994
- [Derived] Blewer AL, Putt ME, McGovern SK, Murray AD, Leary M, Riegel B, Shea JA, Berg RA, Asch DA, Viera AJ, Merchant RM, Nadkarni VM, Abella BS; CHIP Study Group. A pragmatic randomized trial of cardiopulmonary resuscitation training for families of cardiac patients before hospital discharge using a mobile application. Resuscitation. 2020 Jul;152:28-35. doi: 10.1016/j.resuscitation.2020.04.026. Epub 2020 May 3. PMID 32376347
- See also: University of Pennsylvania - Center for Resuscitation Science — https://www.med.upenn.edu/resuscitation/
- See also: American Heart Association — http://www.heart.org/HEARTORG/